CLINICAL TRIAL: NCT05453552
Title: G-CSF+DAC+BUCY vs. G-CSF+DAC+BF Conditioning Regimen for Patients With High-risk MDS Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: G-CSF+DAC+BUCY vs G-CSF+DAC+BF Conditioning Regimen for High-risk MDS Undergoing Allo-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Institute of Hematology & Blood Diseases Hospital, China (Other); Guangzhou First People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First People's Hospital of Chenzhou (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-233
Record Dates: First submitted 2022-07-05; First posted 2022-07-12 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-07

CONDITIONS: Myelodysplastic Syndrome; Allogeneic Hematopoietic Stem Cell Transplantation; Conditioning
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine; Busulfan; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CSF+DAC+BF (Experimental): For patients with high-risk MDS undergoing allo- HSCT, Granulocyte Colony-Stimulating Factor (G-CSF)+Decitabine+BF conditioning regimen was G-CSF 5ug/kg/day on days -17 to -10 (when white blood cell is more than 20G/L, stop using G-CSF), Decitabine 20mg/m2/day on days -14 to -10, Busulfan (BU) 3.2 mg/kg/day on days -6 to -3, Fludarabine (FLU) 30mg/m2/ day on days -7 to -3.
  Interventions: Drug: Granulocyte Colony-Stimulating Factor(G-CSF); Drug: Decitabine (DAC); Drug: Fludarabine (FLU); Drug: Busulfan (BU)
- G-CSF+DAC+BUCY (Active Comparator): For patients with high-risk MDS undergoing allo- HSCT, Granulocyte Colony -Stimulating Factor (G-CSF)+Decitabine+BUCY conditioning regimen was G-CSF 5ug/kg/day on days -17 to -10 (when white blood cell is more than 20G/L, stop using G-CSF), Decitabine 20mg/m2/day on days -14 to -10, Busulfan (BU) 3.2 mg/kg/day on days -7 to -4, Cyclophosphamide (CY) 60 mg/kg/day on days -3, -2.
  Interventions: Drug: Granulocyte Colony-Stimulating Factor(G-CSF); Drug: Decitabine (DAC); Drug: Busulfan; Drug: Cyclophosphamide (CY)

INTERVENTIONS:
Drug: Granulocyte Colony-Stimulating Factor(G-CSF) — G-CSF was administered at 5 ug/kg/day on days-17 to -10. When white blood cell is more than 20G/L, stop using G-CSF.
Drug: Decitabine (DAC) — Decitabine was administered at 20mg/m2/day on days -14 to -10.
Drug: Busulfan — Busulfan was administered at 3.2 mg/kg/day on days -7 to -4 in G-CSF+DAC+BUCY group.
  Arms: G-CSF+DAC+BUCY
Drug: Fludarabine (FLU) — Fludarabine was administered at 30 mg/m2/day on days -7 to -3.
  Arms: G-CSF+DAC+BF
Drug: Cyclophosphamide (CY) — Cyclophosphamide was administered at 60 mg/kg/day on days -3,-2.
  Arms: G-CSF+DAC+BUCY
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days -6 to -3 in G-CSF+DAC +BF group.
  Arms: G-CSF+DAC+BF

SUMMARY:
Allo-HSCT is the most effective way to cure high-risk MDS patients. At present, the best conditioning regimen for high-risk MDS patients undergoing allo-HSCT remains in discussion. In this prospective study, the safety and efficacy of G-CSF+DAC+BUCY and G-CSF+DAC+BF conditioning regimens in high-risk MDS patients undergoing allo-HSCT are evaluated.

DETAILED DESCRIPTION:
Allo-HSCT is the most effective way to cure high-risk MDS patients. At present, the best conditioning regimen for high-risk MDS patients undergoing allo-HSCT remains in discussion. A previous study by the investigators has showed that G-CSF +DAC+BUCY conditioning regimen could reduce the relapse and improve the survival compared with BUCY conditioning regimen, while the two conditioning regimens both have high non-relapse mortality (NRM). Several retrospective and prospective studies have demonstrated that BF conditioning regimen has a lower NRM compared with BUCY conditioning regimen, while the relapse and survival are similar in patients undergoing BF and BUCY conditioning regimens. Based on the above, the investigators design the prospective randomized controlled study to evaluate the safety and efficacy of G-CSF+DAC+BUCY and G-CSF+DAC+BF conditioning regimens in high-risk MDS patients undergoing allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Had a diagnosis of RAEB-1 or RAEB-2 with IPSS-R >3
* Age 18 to 65 years old
* ECOG performance status of 0-2
* HCT-CI of 0-2
* Were willing to undergo allo-HSCT

Exclusion Criteria:

* Therapy-related MDS
* Previous allo-HSCT
* Uncontrolled infections
* Liver or renal dysfunction
* Severe concomitant conditions not suitable for the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Non-relapse mortality (NRM) | 1 year

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year
Disease-free survival (DFS) | 1 year
Cumulative incidence of relapse | 1 year
Adverse effects | within 100 days post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China